CLINICAL TRIAL: NCT03063788
Title: Imaging the HIV Reservoir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: The Peter Doherty Institute for Infection and Immunity (Other); Monash University (Other); Monash Health (Other); Rockefeller University (Other); Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 568/16
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2018-09

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- HIV uninfected (Experimental): A single intravenous infusion of 3mg/kg 3BNC117 combined with Copper-64 to 2 HIV uninfected individuals
  Interventions: Drug: 3BNC117-Copper-64
- HIV infected viremic (Experimental): A single intravenous infusion of 3mg/kg 3BNC117 combined with Copper-64 to 4 HIV infected individuals with viremia who are not receiving antiretroviral therapy
  Interventions: Drug: 3BNC117-Copper-64
- HIV infected aviremic (Experimental): A single intravenous infusion of 3mg/kg 3BNC117 combined with Copper-64 to 4 HIV infected individuals with undetectable HIV viral load who are receiving antiretroviral therapy
  Interventions: Drug: 3BNC117-Copper-64

INTERVENTIONS:
Drug: 3BNC117-Copper-64 — 3 mg/kg 3BNC117 combined with radio-isotope Copper-64

SUMMARY:
Radiolabelling broadly neutralizing anti-HIV antibody 3BNC117 with a Copper-64 radio isotope for infusion into people with HIV followed by MRI/PET scanning to detect HIV in vivo.

DETAILED DESCRIPTION:
This study aims to develop a method to accurately image the size and location of HIV persistence in HIV-infected individuals. The project aims to combine the broadly neutralizing anti-HIV antibody 3BNC117 with a Copper-64 radio isotope for use in a clinical trial.

The clinical trial has three different stages. The first stage is to recruit two HIV uninfected individuals and determine the safety of 3 mg/kg of 3BNC117 combined with Copper-64 and MRI/PET scanning at 1, 24 and 48 hours post infusion. The second stage is to examine the distribution on MRI/PET of the 3BNC117-Copper-64 combination in four HIV-infected individuals with viremia who are not receiving antiretroviral therapy. The final stage is to perform the same intervention in aviremic people with HIV receiving antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria for All Groups:

* Age 18 to 65 years
* Able to give informed consent
* A female, may be eligible to participate if she:
* Is of non-child-bearing potential defined as either post-menopausal or incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
* Is of child-bearing potential with a negative pregnancy test at screening and agrees to use one of the following methods of contraception consistently and for at least 8 weeks after receiving the investigational drug :
* Complete abstinence from 2 weeks prior to investigational drug, and for at least 8 weeks after receiving the investigational drug
* Double barrier method
* Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year
* Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Approved hormonal contraception
* Any other method with published data showing that the expected failure rate is <1% per year

Group specific Inclusion criteria:

Group 1 (HIV-uninfected)

* A negative HIV Ag/Ab test at screening
* Amenable to HIV risk reduction counselling and agrees to maintain behaviour consistent with low risk of HIV exposure

Group 2 (HIV infected viremic off ART)

* Documented HIV-1 infection
* Not on ART for at least 8 weeks with HIV RNA plasma levels between 2,000 - 100,000 copies/ml
* Current CD4+ T cell counts >300 cells/μL
* 3BNC117 sensitivity of subject derived HIV

Group 3 (HIV infected aviremic on ART)

* Documented HIV-1 infection
* Receiving combination ART for at least 12 months
* HIV-1 plasma RNA <50 copies/mL for > 12 months and <20 copies/mL at screening. Episodes of a single HIV plasma RNA 50-500 copies/mL will not exclude participation if the subsequent HIV plasma RNA was <50 copies/mL
* Current CD4+ T cell counts >300 cells/μL

Exclusion Criteria for All Groups:

* Any clinically significant acute or chronic medical condition that in the opinion of the investigator would preclude participation (e.g. lymphoproliferative disorders or significant resections of the gastrointestinal tract that would interfere with the distribution of HIV tissue reservoirs)
* Receipt of a vaccination 14 days prior to receiving investigational drug
* Previous use of histone deacetylase inhibitors or other latency reversing agents
* Receipt of experimental HIV vaccine or monoclonal antibody therapy of any kind in the past
* History of Hepatitis B (Positive HBsAg) or Hepatitis C co-infection (Individuals with prior hepatitis C infection that is now cleared are eligible for enrolment)
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Active alcohol or substance use that in the opinion of the investigator will prevent adequate compliance with study procedures
* Currently pregnant, breastfeeding or unwilling to use barrier contraception
* Women who are pregnant or breastfeeding or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy as specified in the inclusion criteria
* The following laboratory abnormalities:
* Absolute neutrophil count ≤1,300
* Hemoglobin ≤ 10 gm/dL
* Platelet count ≤125,000
* ALT ≥ 2.0 x ULN
* Total bilirubin ≥ 1.5 ULN
* Creatinine ≥ 1.1 x ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Comparisons of PET standard uptake values in regions of interest (gastrointestinal tract, lymph node groups, genital tract, and spleen) between the three groups (uninfected, viremic and aviremic infected) | 2 days
  To determine if there is increased PET uptake in HIV viremic and aviremic groups as compared to uninfected group

SECONDARY OUTCOMES:
Safety and tolerability (adverse events and assessment of laboratory parameters) | 2 weeks
  Reporting of adverse events and assessment of laboratory parameters
Comparisons of PET standard uptake values in regions of interest within each individual to radioactivity levels in a homogenous area of muscle to generate target to muscle ratios. | 2 days
  To determine whether HIV positive participants display organ specific binding of the anti-HIV antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No